CLINICAL TRIAL: NCT01461252
Title: Cryoablation Combined With Radiation Therapy for the Palliation of Painful Bone Metastases
Brief Title: Safety and Efficacy of Cryoablation Combined With Radiation Therapy for the Palliation of Painful Bone Metastases
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients were treated due to enrollment challenges.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CUC10-BNE01
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Pain; Neoplasm Metastasis
Keywords: Painful bone metastases; Bone metastases; Metastatic bone tumors; Metastatic bone pain; Cryoablation; Cryotherapy; Cryosurgery; Radiation therapy; Radiotherapy
MeSH Terms: conditions — Pain; Neoplasm Metastasis; Bone Neoplasms | interventions — Cryosurgery; Cryotherapy; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoablation combined with radiation (Other): All subjects will have cryoablation combined with radiation on one or two painful metastatic bone tumors.
  Interventions: Procedure: Cryoablation; Procedure: Radiation

INTERVENTIONS:
Procedure: Cryoablation — For cryoablation in the palliation of painful bone metastases, subject preparation, anesthesia, intra-operative monitoring, and postoperative management are identical to those of standard cryoablation routinely performed at all clinical centers participating in this study and are at the discretion of the investigator.
  Other Names: Cryotherapy; Cryosurgery; Visual-ICE Cryoabltaion System; SeedNet Cryoablation System; PresIce Cryoablation System; IceRod Cryoablation Needle; IceRod PLUS Cryoablation Needle; IceEDGE 2.4 Cryoablation Needle; IceSeed Cryoablation Needle; IceSphere Cryoablation Needle
Procedure: Radiation — Radiation therapy is usually performed with 6-18 Megavolt photons from a linear accelerator. The proposed dose and frequency of radiation for this protocol are: 8 Gray in 1 fraction, 30 Gray in 10 fractions, or 37.5 Gray in 15 fractions. These proposed doses or other doses will be prescribed at the discretion of the investigator. It is anticipated that subjects will begin the radiation therapy approximately within one to three weeks after the cryoablation procedure. The doses and frequency of the radiation treatment will be collected as well as toxicities.
  Other Names: Radiotherapy

SUMMARY:
This study will evaluate the safety and efficacy of cryoablation therapy combined with radiation therapy for the relief of pain associated with metastatic bone tumors.

DETAILED DESCRIPTION:
Patients with painful bone metastases who meet the eligibility criteria and who have been determined to be an appropriate candidate for cryoablation therapy and radiation therapy will be offered enrollment into the study. Cryoablation is the process of destroying tissue by the application of extremely cold temperatures. Galil Medical Cryoablation Systems are used as a surgical tool in the fields of general surgery, dermatology (skin), neurology (nerves), chest surgery (including lung), Ears-Nose-Throat (ENT), gynecology, oncology (cancer), proctology (colon/rectal) and urology (kidney). Radiation therapy, also called radiotherapy, uses carefully targeted doses of high-energy radiation to kill cancer cells. Radiation is used to treat many kinds of cancer.

Patients agreeing to participate will read and sign an informed consent form and thus become subjects in the study. Treatment will be performed using a Galil Medical cryoablation system and Galil Medical cryoablation needles. Subjects will be followed for up to 24 weeks (6 months) for palliation of pain, quality of life and analgesic usage. Baseline and follow-up data will be collected for each subject via a web-based electronic data collection tool.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Metastatic bone disease with metastatic disease previously confirmed by prior biopsy; or Metastatic bone disease previously confirmed on imaging [e.g. computed tomography (CT) or magnetic resonance imaging (MRI)] with known (biopsied) primary disease (primary bone cancer is excluded)
* Current analgesic therapies have failed OR the subject is experiencing intolerable side effects
* Unremitting pain that resulted in a return visit to the oncologist. The 'worst pain' in the last 24 hours must be reported to be 4 or above on a scale of 0 (no pain) to 10 (pain as bad as subject can imagine) despite pharmaceutical pain management
* Pain must be from one or two painful metastatic sites in the bone that is amenable to cryoablation with CT or MRI (additional less painful metastatic sites may be present)

  • Pain from the reported one or two metastatic sites must correlate with an identifiable tumor on CT, MRI, or ultrasound (US) imaging
* Tumors must be suitable for cryoablation
* If the primary tumor is in the spine, there must be an intact cortex between the mass and the spinal canal and exiting nerve roots
* Cryoablation should be performed within 14 days of baseline evaluations
* Stable use of hormonal therapy (no changes within 4 weeks prior to the cryoablation procedure)
* Stable use of pain medications (no changes within 2 weeks prior to the cryoablation procedure)
* ECOG (Eastern Cooperative Oncology Group) scale performance status 0-3
* Life expectancy ≥ 2 months
* Platelet count >50,000/mm³ within 6 weeks of screening
* INR (International Normalized Ratio) <1.5 within 6 weeks of screening
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up
* If taking antiplatelet or anticoagulation medication, it must be able to be discontinued prior to the procedure for an appropriate amount of time (e.g., aspirin, ibuprofen, low molecular weight heparin preparations)
* Clinically suitable for cryoablation therapy
* Clinically suitable for radiation therapy

Exclusion Criteria:

* Leukemia, lymphoma, and myeloma
* Tumor involves a weight-bearing long bone of the lower extremity with the tumor causing > 50% loss of cortical bone
* Has undergone prior ablation treatment of the index tumor
* Has undergone prior radiation therapy of the index tumor < 3 weeks prior to screening
* Index tumor causing clinical or radiographic evidence of spinal cord or cauda equina compression/effacement
* Anticipated treatment of the index tumor that would require iceball formation within 1.0 cm of the spinal cord, brain, other critical nerve structure, large abdominal vessel such as the aorta or inferior vena cava, bowel, or bladder
* Surgery at the tumor site or surgery involving the cryoablation-treated tumor
* Index tumor involves the skull (treatment of other painful tumors in subjects with skull tumors is not excluded)
* ANC (absolute neutrophil count) <1000 mm3 within 6 weeks of screening
* Uncontrolled coagulopathy or bleeding disorders
* Currently pregnant, nursing, or wishing to become pregnant during the study
* Active, uncontrolled infection
* Serious medical illness, including any of the following: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction, cerebrovascular event within 6 months prior to study entry
* Concurrent participation in other experimental studies that could affect the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Difference in worst pain scores | 24 weeks post cryoablation
  The endpoint for this study will be measured as follows: assessment of the effectiveness of cryoablation combined with radiation associated with palliation of pain in subjects with metastatic bone cancer by measuring the average difference of pre- and posttreatment worst pain in 24 hours from baseline to 24 hour, 1, 4, 12, and 24 week follow-up intervals as measured on the numeric 0 to 10 Brief Pain Inventory (BPI) scale.

SECONDARY OUTCOMES:
Cryoablation retreatments | 24 weeks post-cryoablation
  If the first cryoablation procedure effectively relieves pain but the relief wears off over time and the pain becomes unbearable, a second procedure may be performed. The number of repeat cryoablation treatments will be recorded.
Additional surgical treatments other than cryoablation | 24 weeks post-cryoablation
  If pain is not effectively relieved by the cryoablation, other surgical treatments may be performed. The number of these treatments will be recorded.
Reduced analgesic usage | 24 weeks post-cryoablation
  The number of subjects (percentage) who are able to reduce analgesic medications from baseline to 24 hours, 1, 4, 12, and 24 weeks after cryoablation will be recorded.
Time to maximal palliation of pain after cryoablation | 24 weeks post-cryoablation
  The difference in pain scores will be assessed from baseline to follow-up intervals after cryoablation will be analyzed. The interval indicating the most relief from pain will be compared across subjects.
Number of adverse events | 30 days post-cryoablation
  The safety endpoint for this study is to assess the incidence and severity of intra-operative events, post operative adverse events, serious adverse events and unanticipated adverse device effects related to the cryoablation procedure.
Difference in average pain scores | 24 weeks post-cryoablation
  Difference in average pain scores from baseline to 24 hours, 1, 4, 12, and 24 weeks after cryoablation as measured on the numeric 0 to 10 BPI scale
Time to recurrence of worst pain | 24 weeks post-cryoablation
  Time to recurrence of worst pain at or above baseline; worst pain score in the 24 week follow-up period as measured on the numeric 0 to 10 BPI scale
Subject satisfaction with the amount of palliation of pain obtained from cryoablation combined with radiation | 24 weeks post-cryoablation
  Subject satisfaction will be compared at baseline to follow-up intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Matteo, MD, Study Chair — Shands Medical Center, Jacksonville, FL

REFERENCES:
- [Background] Callstrom MR, Charboneau JW. Image-guided palliation of painful metastases using percutaneous ablation. Tech Vasc Interv Radiol. 2007 Jun;10(2):120-31. doi: 10.1053/j.tvir.2007.09.003. PMID 18070690
- [Background] McQuay HJ, Collins SL, Carroll D, Moore RA. Radiotherapy for the palliation of painful bone metastases. Cochrane Database Syst Rev. 2000;(2):CD001793. doi: 10.1002/14651858.CD001793. PMID 10796822
- [Background] Chow E, Harris K, Fan G, Tsao M, Sze WM. Palliative radiotherapy trials for bone metastases: a systematic review. J Clin Oncol. 2007 Apr 10;25(11):1423-36. doi: 10.1200/JCO.2006.09.5281. PMID 17416863
- [Background] Fairchild A, Barnes E, Ghosh S, Ben-Josef E, Roos D, Hartsell W, Holt T, Wu J, Janjan N, Chow E. International patterns of practice in palliative radiotherapy for painful bone metastases: evidence-based practice? Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1501-10. doi: 10.1016/j.ijrobp.2008.12.084. Epub 2009 May 21. PMID 19464820
- [Background] Callstrom MR, Atwell TD, Charboneau JW, Farrell MA, Goetz MP, Rubin J, Sloan JA, Novotny PJ, Welch TJ, Maus TP, Wong GY, Brown KJ. Painful metastases involving bone: percutaneous image-guided cryoablation--prospective trial interim analysis. Radiology. 2006 Nov;241(2):572-80. doi: 10.1148/radiol.2412051247. PMID 17057075
- [Background] Coleman RE. Management of bone metastases. Oncologist. 2000;5(6):463-70. doi: 10.1634/theoncologist.5-6-463. PMID 11110597
- [Background] Belfiore G, Tedeschi E, Ronza FM, Belfiore MP, Della Volpe T, Zeppetella G, Rotondo A. Radiofrequency ablation of bone metastases induces long-lasting palliation in patients with untreatable cancer. Singapore Med J. 2008 Jul;49(7):565-70. PMID 18695866
- [Background] Simon CJ, Dupuy DE. Percutaneous minimally invasive therapies in the treatment of bone tumors: thermal ablation. Semin Musculoskelet Radiol. 2006 Jun;10(2):137-44. doi: 10.1055/s-2006-939031. Epub 2006 Apr 5. PMID 16598666
- [Background] Ullrick SR, Hebert JJ, Davis KW. Cryoablation in the musculoskeletal system. Curr Probl Diagn Radiol. 2008 Jan-Feb;37(1):39-48. doi: 10.1067/j.cpradiol.2007.05.001. PMID 18054665
- [Background] Hartsell WF, Scott CB, Bruner DW, Scarantino CW, Ivker RA, Roach M 3rd, Suh JH, Demas WF, Movsas B, Petersen IA, Konski AA, Cleeland CS, Janjan NA, DeSilvio M. Randomized trial of short- versus long-course radiotherapy for palliation of painful bone metastases. J Natl Cancer Inst. 2005 Jun 1;97(11):798-804. doi: 10.1093/jnci/dji139. PMID 15928300
- [Background] Wu JS, Wong R, Johnston M, Bezjak A, Whelan T; Cancer Care Ontario Practice Guidelines Initiative Supportive Care Group. Meta-analysis of dose-fractionation radiotherapy trials for the palliation of painful bone metastases. Int J Radiat Oncol Biol Phys. 2003 Mar 1;55(3):594-605. doi: 10.1016/s0360-3016(02)04147-0. PMID 12573746
- [Background] Dupuy DE, Liu D, Hartfeil D, Hanna L, Blume JD, Ahrar K, Lopez R, Safran H, DiPetrillo T. Percutaneous radiofrequency ablation of painful osseous metastases: a multicenter American College of Radiology Imaging Network trial. Cancer. 2010 Feb 15;116(4):989-97. doi: 10.1002/cncr.24837. PMID 20041484
- [Background] Callstrom MR, York JD, Gaba RC, Gemmete JJ, Gervais DA, Millward SF, Brown DB, Dupuy D, Goldberg SN, Kundu S, Rose SC, Thomas JJ, Cardella JF; Technology Assessment Committee of Society of Interventional Radiology. Research reporting standards for image-guided ablation of bone and soft tissue tumors. J Vasc Interv Radiol. 2009 Dec;20(12):1527-40. doi: 10.1016/j.jvir.2009.08.009. Epub 2009 Oct 27. No abstract available. PMID 19864161